CLINICAL TRIAL: NCT02283346
Title: Single Fraction High Dose Rate (HDR) Brachytherapy Plus Hypofractionated External Beam Radiotherapy (EBRT) for Low-risk Prostate Cancer: Phase II Trial
Brief Title: Single Fraction HDR Brachytherapy Plus Hypofractionated EBRT for Low-risk Prostate Cancer: Phase II Trial
Acronym: AC-P01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-P01
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; HDR brachytherapy; hypo fractionated external beam radiotherapy; toxicity; biochemical control
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HDR Brachytherapy + EBRT (Experimental): HDR brachytherapy + hypofractionated EBRT
  Interventions: Radiation: HDR brachytherapy + hypofractionated EBRT

INTERVENTIONS:
Radiation: HDR brachytherapy + hypofractionated EBRT — Single Fraction High Dose Rate (HDR) Brachytherapy One fraction with 10-15 Gray (Gy) (depending on normal tissues constraints).
  + Hypofractionated External Beam Radiotherapy (EBRT) The treatment will be held with fractions 2.5 Gy per day, with a final dose between 25 and 50 Gy (depending on normal tissues constraints).

SUMMARY:
The hypofractionated external radiation (EBRT) is a technique that radiation dose delivery using higher daily fractions than those used routinely. In this way can cause more damage tumor, especially in tissues that have a slower proliferation rate, as in the case of prostate cancer. Furthermore, achieves a reduction in total treatment time and probably a lesser chance of development of collateral in tissues of high multiplication rate as the lining of the rectum and bladder effects.

With brachytherapy boost for high dose rate is achieved by administering a more intense dose on the tumor and lower the sound around the region to be treated tissues, improving the therapeutic window.

Treatment with retracted and fully ambulatory time, has potential benefit as early patient return to usual activities and optimizing the flow of patients who require treatment with radiotherapy. This prospective study aims to assess the results and the toxicity profile of this treatment regimen retracted.

DETAILED DESCRIPTION:
OBJECTIVE The primary objective is to analyze the toxicity profile, via a phase II study of treatment of patients with low risk prostate cancer with the association of hypo fractionated EBRT and HDR brachytherapy boost.

It will also analyze the biochemical control and expense to the procedure.

STUDY DESIGN Prospective phase II study and not randomized. Patients with localized low-risk prostate cancer will be recruited to participate in protocol hypofractionated external beam radiotherapy followed by brachytherapy high dose rate.

INCLUSION CRITERIA

* Biopsy confirming adenocarcinoma of the prostate;
* Low risk prostate cancer: less than or equal T2a, and less than or equal to 10 ng PSA / ml stage and Gleason score less than or equal to 6
* Prostate volume less than or equal to 60cc.

EXCLUSION CRITERIA

* Patients under 18 or over 90 years;
* Adjuvant Hormone (any duration);
* Prior pelvic radiotherapy;
* Adjuvant Chemotherapy.

OUTCOMES

Primary outcomes:

Reduction of rectal acute morbidity (within three months of treatment) and late (after three months to twelve months from the last treatment recruited patient).

Reduction of acute urinary morbidity (within three months of treatment) and late (after three months to twelve months from the last treatment recruited patient).

The primary outcomes (toxicity) will be evaluated in patients who receive more than 90% of the intended dose protocol with crte and HDR brachytherapy.

(Scale used: CTCAE v4.03, Published online: May 28,2009 by the United States Department of Health and Human Services - NIH - attached).

Secondary outcomes:

Biochemical control (serial PSA measurements at intervals of three months in the first year, four months in the second year, six months of the third year onwards).

Cost-analysis procedure

STAGING

Performing the following tests:

1. Physical examination - rectal (TR)
2. transrectal US (TRUS)
3. pelvic CT
4. serum prostatic specific antigen (PSA) dosage
5. Bone Scan

ETHICAL ASPECTS The treatment regimen will be monitored for the possible emergence of excessive toxicity, considering that the same appearance in more than 25% of cases will be cause for termination of the protocol.

The study will begin after approval by the Research Ethics Committee (CEP) of the AC Camargo Cancer Center. Each patient will sign a term of informed consent (IC) prior to study entry. The term was written in accessible layman's language the patient, following the ethical recommendations. Patients may withdraw from the study at any time, without prejudice to the proposed treatment. We declare the confidentiality of personally identifiable patient, it is not possible to identify it during analysis and publication of data.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirming adenocarcinoma of the prostate
* Low-risk Prostate Cancer: less than or equal T2a stage + PSA less than or equal to 10 ng/ml stage + Gleason score less than or equal to 6
* Prostate volume than or equal to 60cc

Exclusion Criteria:

* Adjuvant Hormone
* Prior pelvic radiotherapy
* Adjuvant Chemotherapy

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Acute and Late rectal and urinary morbidity | 12 weeks
  toxicity associated with the rectum and urinary tract, using Common Terminology Criteria for Adverse Events v4.0 (CTCAE v4.0)

SECONDARY OUTCOMES:
biochemical control | 3 years
  serum PSA increase (2.0ng/ml above the nadir)
costs analysis of the treatment | one week after the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lucas G Sapienza, MD, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil